CLINICAL TRIAL: NCT06467552
Title: Effects of Nutritional Support on Postoperative Delirium (POD) in Elderly Non-cardiac Surgical patients_non-inferiority Comparison
Brief Title: Effects of Nutritional Support on Postoperative Delirium
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 4-2024-0324
Record Dates: First submitted 2024-05-20; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-05

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): The entire process is carried out according to Severance Hospital surgical protocols.
  Interventions: Procedure: control group
- intervention group (Experimental): The entire process is carried out according to Severance Hospital surgical protocols. The patients of control group will receive education from the research team about the importance of nutrition and exercise before and after surgery. In addition, the patients of control group will be instructed to take up to 4 doses of the nutritional supplement (Nucare Curact provided by DAESANG Wellife Inc.) per day for approximately 2 weeks before surgery and for about 4 weeks after surgery.
  Interventions: Dietary Supplement: Nucare Curact group

INTERVENTIONS:
Procedure: control group — The entire process is carried out according to Severance Hospital surgical protocols.
  Arms: control group
Dietary Supplement: Nucare Curact group — The entire process is carried out according to Severance Hospital surgical protocols. The patients of control group will receive education from the research team about the importance of nutrition and exercise before and after surgery. In addition, the patients of control group will be instructed to take up to 4 doses of the nutritional supplement (Nucare Curact provided by DAESANG Wellife Inc.) per day for approximately 2 weeks before surgery and for about 4 weeks after surgery.
  Arms: intervention group

SUMMARY:
This study is a prospective, single-center, randomized controlled trial to compare whether applying nutritional supplementation therapy before and after surgery in elderly patients aged 65 years or older undergoing non-cardiac surgery can reduce the incidence of postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients aged 65 and above.
* Patients undergoing non-cardiac major surgery in thoracic surgery, lung cancer surgery, multi-level spinal surgery in neurosurgery and orthopedics, or liver cancer surgery in hepatobiliary and pancreatic surgery, under general anesthesia with an expected surgery duration of 2 hours or more.
* Patients scheduled for arterial catheterization.
* Patients who are able to take oral intake from postoperative day #1.

Exclusion Criteria:

* Patients with uncontrolled systemic conditions such as diabetes, hypertension, renal disease, liver disease, and other systemic illnesses.
* Those with visual impairment.
* Patients with cognitive impairment based on the Mini-Mental State Examination for Dementia Screening criteria.
* Individuals experiencing difficulty in communication.
* Those diagnosed with neurological disorders (such as brain hemorrhage, stroke, brain tumor, dementia, Parkinson's disease, cognitive impairment, depression, etc.).
* Patients diagnosed with alcohol or substance addiction.
* Patients with cancelled scheduled surgeries.
* Patients undergoing minor surgeries with expected anesthesia durations of less than 2 hours.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2028-05-12 (Estimated); Study Completion 2028-05-12 (Estimated)

PRIMARY OUTCOMES:
incidence of postoperative delirium | from postoperative day 0 to postoperative day 7
  Confusion assessment methods(CAM) will be used for diagnosing delirium At least two times a day during the hospitalization period. Patients diagnosed with delirium using the CAM were evaluated for the duration, symptoms, and type of delirium (e.g., reduced awareness of the environment; poor cognitive skills; behavioral changes; and emotional disturbances).
  ** Confusion assessment methods(CAM) diagnostic algorism (positive or negative result, positive means delirium)
  CAM is considered positive if features 1 and 2 are present, with at least one of features 3 or 4. Below are the four criteria of features :
  1. Acute onset and fluctuating course Determined by collateral history or repeated clinic assessment
  2. Inattention Counting from 20-1 is a simple (if blunt) test for this
  3. Disorganized thinking
  4. Altered levels of consciousness

SECONDARY OUTCOMES:
duration of delirium | from postoperative day 0 to postoperative day 7
  The Quality of Recovery-40 (QoR-40) : 40~200(better recovery)
type of delirium | from postoperative day 0 to postoperative day 7
K-FRAIL for frailty | from postoperative day 0 to postoperative day 7
  The Korean version of the fatigue, resistance, ambulation, illnesses, and loss of weight (K-FRAIL) scale : 0(healthy)~8(frail).
  A raw score is standardized. A lower score means cognitive dysfunction.
GDS for depression | from postoperative day 0 to postoperative day 7
  Geriatric Depression Scale(GDS) : 0(normal)~ 15(depression). A raw score is standardized. A lower score means cognitive dysfunction.
ADL for independence | from postoperative day 0 to postoperative day 7
  Activities of Daily Living(ADL)-Barthel Index : 0(completely dependent )~105( independent).
  A raw score is standardized. A lower score means cognitive dysfunction.
SNSB-c for cognitive dysfunction | from postoperative day 0 to postoperative day 7
  Seoul Neuropsychological Screening Battery-Core(SNSB-C): total score is 617. A raw score is standardized. A lower score means cognitive dysfunction.
QOR-40 for recovery | from postoperative day 0 to postoperative day 7
  The Quality of Recovery-40 (QoR-40) : 40~200(better recovery)
K-MoCA for cognitive dysfunction | from postoperative day 0 to postoperative day 7
  Korean-Montreal Cognitive Assessment(K-MoCA) : 0~30, cognitive dysfunction<23.
IADL for independence | from postoperative day 0 to postoperative day 7
  Instrumental Activities of Daily Living(IADL)-Lawton-Brody Scale : 0~8(complete independence).

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health system, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No